CLINICAL TRIAL: NCT01335893
Title: A Phase 1, Open-Label, Single Center Study of the Imaging Potential of Indocyanine Green in Subjects Undergoing Thoracic Surgery Presenting With Lung Nodules
Brief Title: Intraoperative Imaging of Thoracic Malignancies With Indocyanine Green
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UPCC:11510
Record Dates: First submitted 2011-04-01; First posted 2011-04-14 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Lung Neoplasms
Keywords: Imaging; Indocyanine Green; Lung Cancer; Lung Neoplasms; Preliminary Study
MeSH Terms: conditions — Lung Neoplasms | interventions — Indocyanine Green; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ICG injection group (Experimental): This group will receive a single dose of ICG, diluted in saline solution, prior to surgery. Then, during their surgery, they will be imaged with the camera and imaging probe we have developed.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Dose will be diluted in saline solution. This will be a single dose given before the surgery intravenously.
  Other Names: ICG; Indocyanine Green USP, for injection

SUMMARY:
Our specific aim is to determine if Indocyanine Green (ICG) administered intraoperatively and imaged using our camera will aid in the identification of a suspected lung nodule.

DETAILED DESCRIPTION:
According to the World Health Organization, lung cancer is the most common cause of cancer-related death in men and women, and is responsible for 1.3 million deaths worldwide annually as of 2004. Surgery remains the best option for patients presenting with operable Stage I or II cancers, however the five year survival rate for these candidates remains at a dismal 53% for Stage I and 32% for Stage II1. The high rates of recurrence suggest that surgeons are unable to completely detect and remove primary tumor nodules in a satisfactory manner as well as lingering metastases in sentinel lymph nodes. By ensuring a negative margin through near-infrared imagery with a safe non-toxic contrast agent it would be possible for the investigators to improve the rates of recurrence free patients and thus overall survival. This study is a small pilot/feasibility study to determine if the investigators camera system can be effective at identifying malignancies in lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over 18 years of age
2. Patients presenting with a lung nodule or mass presumed to be resectable stage I, II, or IIIa non-small call lung cancer on pre-operative assessment
3. Good operative candidate as determined by a thoracic oncology multidisciplinary team
4. Subject capable of giving informed consent and participating in the process of consent

Exclusion Criteria:

1. Pregnant women as determined by urinary or serum beta hCG within 72 hours of surgery
2. Subjects with a history of iodide allergies
3. At-risk patient populations

   * Homeless patients
   * Patients with drug or alcohol dependence
   * Children and neonates
   * Patients unable to participate in the consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12-14 (Actual)

PRIMARY OUTCOMES:
Imaging effectiveness of ICG and imaging system. | 1 day after injection of ICG
  The primary end-point of the study is to determine the sensitivity of ICG uptake and expression in identifying lung nodules / masses when excited by an imaging probe intraoperatively. This will be accomplished by using the probe to image the tumor, then subtracting the background from surrounding thoracic structures. Uptake will be measured using the scale of the instrument, an arbitrary value of between 1 and 10,000. Uptake will be summarized using the mean and 95% confidence interval (CI).

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Singhal, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Okusanya OT, Holt D, Heitjan D, Deshpande C, Venegas O, Jiang J, Judy R, DeJesus E, Madajewski B, Oh K, Wang M, Albelda SM, Nie S, Singhal S. Intraoperative near-infrared imaging can identify pulmonary nodules. Ann Thorac Surg. 2014 Oct;98(4):1223-30. doi: 10.1016/j.athoracsur.2014.05.026. Epub 2014 Aug 5. PMID 25106680